CLINICAL TRIAL: NCT01953224
Title: STEP AND GO: A Study of Technology-based Exercise Promotion and Gaming Outcomes
Brief Title: STEP AND GO: A Study of Technology-based Exercise Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-0285
Record Dates: First submitted 2013-09-06; First posted 2013-09-30 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-04

CONDITIONS: Cardiovascular Disease; Obesity; Cancer; Diabetes
Keywords: Physical activity; Video game; Mobile; Technology; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Neoplasms; Diabetes Mellitus; Motor Activity | interventions — Jogging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Game-based intervention (Experimental): This arm will receive the game intervention, which will include provision of a mobile smartphone device, cellular data service, the game application loaded onto the device, credit to load approximately 40-50 songs onto the device, headphones, and an armband for wearing the device. Participants will also receive weekly counseling calls.
  Interventions: Behavioral: Game-based intervention; Device: Smartphone
- Wait list control (No Intervention): This group will receive no intervention until after completion of the final assessment of the randomized trial. Then, they will receive the full intervention.

INTERVENTIONS:
Behavioral: Game-based intervention — Investigators will provide participants with a smartphone and required accessories (gift card for downloading the game application and music, headphones, armband). The game, "Zombies, Run!" encourages walking/jogging by playing music interspersed with a continuous narrative. Periodic "zombie chases" encourage brief interval training. Participants will set goals to increase their activity and receive weekly brief counseling phone calls to provide feedback.
  Other Names: Zombies, Run!
  Arms: Game-based intervention
Device: Smartphone
  Arms: Game-based intervention

SUMMARY:
The purpose of the study is to test an intervention that uses a mobile game to encourage increased physical activity among adults.

DETAILED DESCRIPTION:
Physical activity reduces cardiometabolic risk factors. Unfortunately, a majority of adults do not meet activity recommendations. Though walking is a preferred method for activity with proven effectiveness, motivating sustained adherence to activity goals is difficult. "Gamification" using technology-based tools holds promise for motivating increased adherence to physical activity goals. Gamification occurs when elements from video games (such as leaderboards, badges, and progression through a virtual narrative) are integrated into non-game applications. Game elements may motivate faster, longer, and/or more frequent walking by making walking and self-monitoring more enjoyable. In the proposed research the investigators seek to test the feasibility and acceptability of a technology-based intervention that "gamifies" physical activity using technology. The investigators will randomize 40 inactive overweight adults (20 women, aged 18 - 69) to either an intervention group or a wait-list control. (Note: 10 additional participants will be recruited for a pre-pilot one-arm test of the intervention to ensure that the mobile devices, cellular service, game, etc. are working correctly.) The intervention will consist primarily of provision of a mobile device loaded with a narrative-based walking application ("app"). Participants will be instructed to use the app to achieve activity goals increasing from 60 to 150 or more minutes per week. The app uses global positioning systems and accelerometry to track exercise duration and intensity. Investigators will call participants weekly for brief counseling and technical support. The intervention will last 12 weeks. Primary outcomes are process measures of feasibility and acceptability, including attrition, reasons for drop-out, adherence to use of the app, exposure to calls, and any adverse events. The investigators will also compare behavioral (physical activity), weight-related (weight, body composition), and health outcomes (fitness, blood pressure) in the intervention group to the wait-list control. Finally, theory-based intermediate variables, such as self-efficacy, intrinsic motivation, and self-regulation, will also be investigated. This study will provide crucial information regarding the promise of gamified apps and will lay a foundation for a larger research program in technology-based cardiovascular health promotion.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 69 years old
2. BMI is between 25 kg/m2 and 35 kg/m2
3. Able to read and understand English
4. Able to read words in standard applications on a mobile device 5" large
5. Able to walk for exercise
6. Able to find transportation to the study location
7. Willing to use a smartphone provided by the study to participate
8. Willing to listen to a potentially scary or sad story that includes violence
9. Willing to share basic information on walks with other participants via a social network

Exclusion Criteria:

1. (If female) currently pregnant or nursing or plan to become pregnant in the next 6 months
2. Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q, items 1 - 4). Reporting taking medicine for blood pressure on this questionnaire will require a doctor's note to participate.
3. Unable to walk for exercise (self-report)
4. Report current symptoms of alcohol or substance dependence
5. Plans to move away from the Galveston-Houston area in the next 4 months or to be out of town for more than 1 week during the study period
6. Unwillingness to report drugs taken for comorbidities such as hypertension or diabetes
7. Takes medications for diabetes or thyroid issues
8. Stroke, hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
9. Participant is active (60 minutes of moderate-vigorous intensity activity per week or more)
10. Another member of the household is a participant or staff member on this trial
11. Currently a participant in a physical activity or weight loss research trial
12. Recently (less than six months ago) completed a physical activity or weight loss research trial
13. Recently (less than six months ago) lost more than 5% of their body weight
14. Report a history of orthopedic complications that would prevent optimal participation in the physical activities prescribed (e.g., heel spurs, severe arthritis - may be eligible, but a doctor's note will be required)
15. Current smoker
16. Currently uses Zombies, Run! for exercise

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Lyons, PhD, MPH, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-pilot results (N = 10) are not reported here, as outcomes are not comparable to those from the main trial. Specifically, the pre-pilot tested assignment of mobile phones to individuals as a delivery method for the intervention, which was found to be not feasible. Conclusions from the pre-pilot about intervention content would be biased.
Groups:
- Game-based Intervention: This arm will receive the game intervention, which will include provision of a mobile smartphone device, cellular data service, the game application loaded onto the device, credit to load approximately 40-50 songs onto the device, headphones, and an armband for wearing the device. Participants will also receive weekly counseling calls.
  Game-based intervention: Investigators will provide participants with a smartphone and required accessories (gift card for downloading the game application and music, headphones, armband). The game, "Zombies, Run!" encourages walking/jogging by playing music interspersed with a continuous narrative. Periodic "zombie chases" encourage brief interval training. Participants will set goals to increase their activity and receive weekly brief counseling phone calls to provide feedback.
  Smartphone
Period: Overall Study
Arm/Group | Game-based Intervention | Wait List Control
Started | 20 | 20
Completed | 18 | 17
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Game-based Intervention | Wait List Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (13.44) | 49.1 (12.01) | 48.00 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity From Baseline to 12 Weeks
Description: Minutes of physical activity measured over a 7 day period. Baseline values were carried forward for participants lost to followup.
Time Frame: Baseline to 12 weeks
Population: Four participants' baseline data were found to be invalid based on standard protocols for accelerometer data cleaning/preparation (i.e., 4 days of 10+ hours wear time)
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Game-based Intervention | Wait List Control
Number analyzed (Participants) | 18 | 18
minutes per day | 8.82 (19.24) | 2.32 (17.13)

2. Secondary Outcome: Change in Physical Fitness From Baseline to 12 Weeks
Description: Maximal treadmill test to measure fitness (operationalized as the amount of oxygen used by the body during maximal effort). Baseline values were carried forward for participants lost to followup.
Time Frame: Baseline to 12 weeks
Population: Several participants did not provide usable data at baseline due to feasibility issues with our measurement protocols. Their data were not included here.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Game-based Intervention | Wait List Control
Number analyzed (Participants) | 15 | 14
mL/kg/min | -0.01 (1.63) | 0.15 (1.32)

3. Secondary Outcome: Change in Body Fat Percentage From Baseline to 12 Weeks
Description: We will use dual x-ray absorptiometry to measure body fat percentage. Baseline values were carried forward for participants lost to followup.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percent body fat
Arm/Group | Game-based Intervention | Wait List Control
Number analyzed (Participants) | 20 | 20
percent body fat | -0.41 (1.00) | -0.20 (1.33)

4. Secondary Outcome: Change in Blood Pressure From Baseline to 12 Weeks
Description: Systolic and diastolic blood pressure will be measured using standard methods. Baseline values were carried forward for participants lost to followup.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Game-based Intervention | Wait List Control
Number analyzed (Participants) | 13 | 16
mmHg
  systolic | 3.62 (9.83) | 2.44 (8.37)
  diastolic | 0.42 (7.84) | -0.88 (2.80)

5. Secondary Outcome: Change in Weight From Baseline to 12 Weeks
Description: We will measure weight using a calibrated scale. Baseline values were carried forward for participants lost to followup.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Game-based Intervention | Wait List Control
Number analyzed (Participants) | 20 | 20
pounds | 0.02 (2.01) | -0.18 (2.44)

6. Secondary Outcome: Change in Motivation From Baseline to 12 Weeks
Description: We will measure intrinsic motivation using the intrinsic regulation subscale from the Behavioral Regulation in Exercise Questionnaire-2. This measure uses a scale from 0 (not true for me) to 4 (very true for me). Positive changes indicate increases in intrinsic motivation over time. Baseline values were carried forward for participants lost to followup.
Time Frame: Baseline to 12 weeks
Population: One participant did not provide usable data at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Game-based Intervention | Wait List Control
Number analyzed (Participants) | 20 | 19
units on a scale | 0.76 (0.97) | 0.18 (0.73)

7. Other Pre Specified Outcome: Number of Participants Who Drop Out of the Study From Baseline to 12 Weeks
Description: We will investigate the number of participants who drop out of the intervention group in comparison to the control group and to norms for similar studies
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Acceptability
Description: Acceptability will be self-reported using a variety of items taken from previous studies of physical activity interventions and usability
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Frequency of App Use Over 12 Weeks
Description: Based on objective measures taken from individual game accounts, we will determine the discrete number of uses of the game app
Time Frame: 12 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Number of Counseling Calls Completed From Baseline to 12 Weeks
Description: Based on counselor logs, we will determine the number of counseling phone calls completed for each participant
Time Frame: 12 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: We will inquire about potential adverse events during counseling calls and assessment visits. Discrete events will be summed, and the number of participants with events will be summed.
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse event information was collected systematically during weekly phone calls and assessments based on a standard protocol.
Arm/Group | Game-based Intervention | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Game-based Intervention (N=20) | Wait List Control (N=20)
Acid reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
strep throat (Infections and infestations) | 0 (0) | 1 (1)
injury to jaw (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
migraine (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a pilot/feasibility study. Sample sizes for the maximal fitness tests and blood pressure were low due to difficulties with feasibility for those measures. Analyses used the intent to treat principle.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No